CLINICAL TRIAL: NCT01105845
Title: Genetics of Motor Learning
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100092; 10-N-0092
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2015-12-21

CONDITIONS: Parkinson s Disease; Dystonic Disorders; Focal Dystonia; Movement Disorders
Keywords: Motor Learning; Genetic Analysis; BDNF; Parkinson Disease; Movement Disorders; Dystonia; Healthy Volunteer; HV
MeSH Terms: conditions — Parkinson Disease; Dystonic Disorders; Movement Disorders; Dystonia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- New studies in human genetics have revealed information about genetic connections to memory and motor behavior. Researchers are interested in investigating the role of genetics in motor learning, in conjunction with related studies taking place in the Human Motor Control Section of the National Institute of Neurological Diseases and Stroke (NINDS). Participants in motor learning studies conducted at NINDS will be asked to provide blood samples for further evaluation.

Objectives:

- To create a repository of blood samples from patients and healthy subjects who are participating in NINDS motor learning studies.

Eligibility:

- Individuals between 18 and 100 years of age who are or will be participating in motor learning research studies at the National Institutes of Health.

Design:

* Blood draws for genetic testing will usually be done on the same day as the motor learning study. Participants will provide one blood sample for research.
* No treatment will be provided under this study....

DETAILED DESCRIPTION:
OBJECTIVE:<TAB>

The objective of this study is to create a bio-repository of blood samples from patients and healthy subjects who are participating in NINDS motor learning studies. Blood will be analyzed for BDNF and samples stored for future genetic studies. . A variety of genes that may affect motor learning are being increasingly identified, and variations among these genes, referred to as polymorphisms, may help explain individual differences.

STUDY POPULATION: <TAB>

We will enroll up to five hundred healthy volunteers and five hundred volunteers with movement difficulties who are between the ages of 18 and 100 and who are already participating, or will be participating, in other protocols dealing with motor learning research studies at the National Institutes of Health (NIH).

DESIGN:<TAB>

This is an observational and repository protocol that involves a single blood sample for genetic analysis. This will allow the genetic characterization of subjects participating in motor learning protocols to be analyzed and tested for the role of genetics in motor learning results.

OUTCOME MEASURE:

We will compare genetic variations with the different behavioral, electrophysiologic, imaging, or other outcomes acquired in the associated motor learning studies. Thus, we will determine whether specific polymorphisms are associated with different measures of motor learning.

ELIGIBILITY:
* INCLUSION CRITERIA:

<TAB>

Anyone aged 18-100 years and participating in a motor learning study at NIH is eligible to participate in this study.

<TAB>

EXCLUSION CRITERIA:

Anyone with impaired decisional capacity, inability to provide informed consent, or who is unable to safely give blood is not eligible to participate in this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-04-14; Study Completion 2015-12-21

PRIMARY OUTCOMES:
Genetic polymorphism frequency (e.g. BNDF Va166Met) compared to measures of motor learning (e.g. reaction time or fMRI BOLD signal change)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Brunoni AR, Lopes M, Fregni F. A systematic review and meta-analysis of clinical studies on major depression and BDNF levels: implications for the role of neuroplasticity in depression. Int J Neuropsychopharmacol. 2008 Dec;11(8):1169-80. doi: 10.1017/S1461145708009309. Epub 2008 Aug 28. PMID 18752720
- [Background] Cheeran B, Talelli P, Mori F, Koch G, Suppa A, Edwards M, Houlden H, Bhatia K, Greenwood R, Rothwell JC. A common polymorphism in the brain-derived neurotrophic factor gene (BDNF) modulates human cortical plasticity and the response to rTMS. J Physiol. 2008 Dec 1;586(23):5717-25. doi: 10.1113/jphysiol.2008.159905. Epub 2008 Oct 9. PMID 18845611
- [Background] Egan MF, Kojima M, Callicott JH, Goldberg TE, Kolachana BS, Bertolino A, Zaitsev E, Gold B, Goldman D, Dean M, Lu B, Weinberger DR. The BDNF val66met polymorphism affects activity-dependent secretion of BDNF and human memory and hippocampal function. Cell. 2003 Jan 24;112(2):257-69. doi: 10.1016/s0092-8674(03)00035-7. PMID 12553913